CLINICAL TRIAL: NCT04087980
Title: Multicenter Pilot Study of the Poseidon System for the Ablation of Prostate Tissue Utilizing Sterile Water Vapor in Patients With Intermediate Risk Localized Prostate Cancer
Brief Title: Ablation of Prostate Tissue Utilizing Sterile Water Vapor in Patients With Intermediate Risk Localized Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francis Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAPOR I Pilot Study
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Poseidon System Treatment (Experimental)
  Interventions: Device: Poseidon System

INTERVENTIONS:
Device: Poseidon System — Multicenter Pilot Study of the Poseidon System for the Ablation of Prostate Tissue Utilizing Sterile Water Vapor in Patients with Intermediate Risk Localized Prostate Cancer

SUMMARY:
The purpose of this research study is to collect information on a new treatment of prostate tissue participants with intermediate risk prostate cancer using a medical device called the Poseidon System. The Poseidon System is intended to ablate prostate tissue in areas of the prostate where cancer has been identified. The medical device delivers thermal energy in the form of water vapor to the prostate tissue through the urethra. Previous research has shown successful prostate tissue ablation. Additional research may help show successful ablation of the prostate tissue where cancer is located.

ELIGIBILITY:
Inclusion Criteria:

* 45-80 years old
* Biopsy confirmed unilateral, adenocarcinoma of the prostate
* Minimum of 12 biopsy cores obtained ≥4 weeks and ≤12 months before treatment. Targeted fusion biopsy is preferred if there is a MRI PI-RADs ≥3 lesion. It is preferred a standard 12 sector biopsy is mapped. MRI required if biopsy was completed >6 months prior to treatment date to confirm no MRI progression of disease that would be considered exclusionary.
* ≤4 of 6 standard sector biopsy cores positive for prostate cancer (unilateral); positive core(s) from a targeted lesion count as one positive core.
* Gleason score of 7 (3+4) / International Society of Urological Pathologists (ISUP) Gleason Grade Group (GGG) 2
* Clinical Stage less than or equal to T2b N0 M0
* PSA (Prostate Specific Antigen) less than or equal to 15ng/mL
* Prostate size 20-80cc

Exclusion Criteria:

* Malignant tumors identified by extraprostatic extension, sphincter involvement/lesion abutment seminal vesicle invasion or lymph node invasion or metastasis
* Narrow Peripheral Zone
* MRI identified PI-RADs ≥4 lesion contralateral to the side that has biopsy confirmed adenocarcinoma
* Prior definitive treatment of prostate cancer

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Serious device related adverse events | 180-day follow-up

SECONDARY OUTCOMES:
Adverse events, serious and non-serious, related and unrelated, will be collected on all patients enrolled | Up to 1 Years
Changes from baseline in the Expanded Prostate Cancer Index Questionnaire (EPIC) | 180-day follow-up
Changes from baseline in the International Index of Erectile Function Questionnaire (IIEF) | 180-day follow-up
Changes from baseline in the International Prostate Cancer Symptom Score (IPSS) | 180-day follow-up
Changes from baseline in the Male Sexual Health Ejaculatory Function Short Form Questionnaire (MSHQ-EjD) | 180-day follow-up
Participants evaluated for Gleason pattern 4 or higher disease on the treated side identified from biopsy | 180-day follow-up
Participants evaluated for biopsy negative on the treated side | 180-day follow-up
Changes from baseline with the PSA (Prostate Specific Antigen) | Up to 1 Year
Changes from baseline with the size of the prostate via MRI (Magnetic Resonance Imaging) | 180-day follow-up
Participants evaluated for Gleason pattern 4 or higher disease on the contralateral side identified from biopsy | 180-day follow-up
Participants evaluated for biopsy negative on the contralateral side | 180-day follow-up

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Chesapeake Urology, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Minnesota Urology, Woodbury, Minnesota
  - Bon Secours/Good Samaritan Hospital, New York, New York
  - Urology San Antonio, San Antonio, Texas